CLINICAL TRIAL: NCT01039142
Title: EFFICACY AND SAFETY OF ACITRETIN IN DOSES OF 25mg,35mg or50mg IN PATIENTS WITH SEVERE PLAQUE TYPE PSORIASIS: A RANDOMISED,DOUBLE BLIND , PARALLEL GROUP DOSE- RANGING STUDY
Brief Title: Dose Ranging Study to Assess the Efficacy and Safety of Acitretin in Severe Plaque Type Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Dr Aklish Jain, Postgraduate Institute of Medical Education and Research
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12345
Record Dates: First submitted 2009-12-23; First posted 2009-12-24 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2008-02

CONDITIONS: Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Acitretin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 25 mg acitretin (Active Comparator): capsule acitretin 25 mg/day will be administered to each patient for a period of 12 weeks
  Interventions: Drug: Acitretin
- 35 mg acitretin (Active Comparator): capsule acitretin 35 mg/day will be administered to each patient for a period of 12 weeks
  Interventions: Drug: Acitretin
- 50 mg acitretin (Active Comparator): capsule acitretin 50 mg/day will be administered to each patient for a period of 12 weeks
  Interventions: Drug: Acitretin

INTERVENTIONS:
Drug: Acitretin — capsule acitretin in dose of 25 mg, 35 mg or 50 mg/ day for 12 weeks or reduction in PASI score by 75% whichever is earlier

SUMMARY:
In this study, the investigators will intend to compare the efficacy and safety of various doses of acitretin in a randomized double blind manner in patients with severe plaque-type psoriasis, by i) studying the change PASI score from baseline as a measure of efficacy ii) determining the frequency of side effects at various doses. Sixty patients will be recruited from Psoriasis Clinic of Department of Dermatology, Venerology and Leprology, PGIMER. Patients will be randomly assigned to one of the three groups: Group A, consisting of 20 patients, will be administered acitretin 25 mg/ day ,Group B, consisting of 20 patients, will be administered acitretin 35 mg/day and GROUP C consisting of 20 patients, will be administered acitretin 50 mg/day This therapy will be continued until PSORIASIS AREA AND SEVERITY INDEX (PASI) scores are reduced to < 25% of the original scores or 12 weeks, whichever comes earlier. It is expected that acitretin at higher doses will be more efficacious . As the exact etiopathogenesis of psoriasis is not fully known, it is difficult to provide a definite cure to all patients, though the disease activity can be controlled to a great extent with various treatment modalities. However the dosage of acitretin be adjusted according to response of the patients and tolerability of side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with plaque-type psoriasis having <90%of body surface area involvement, whose disease activity had been stable for the last 1month.
* Age range 18-65 years of either sex
* Females who are postmenopausal or tubectomised or have completed their family and are willing to maintain contraception 1 month before, during and 2 years after completion of treatment and negative pregnancy tests within 2 months of starting of treatment.
* Compliance for scheduled visit.

Exclusion Criteria:

* Patients with severe hepatic, renal or other systemic disorders (serum bilirubin,AST,ALT and alkaline phosphatase>1.5 times upper limit of normal;serum creatinine >1.5 mg% in males and >1.4mg% in females)
* Pregnant or lactating women,contemplating pregnancy in next 2 -3 years
* Alcoholic
* Metabolic disorders such as hyperlipidemia
* Obese/BMI≥ 30 kg/m2
* Ischemic heart diseases,neuropsychiatric illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-03; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Change in Psoriasis area severity index from baseline to 12 weeks after acitretin therapy | 12 weeks

SECONDARY OUTCOMES:
Frequency of adverse effects at 3 different doses of acitretin | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Dogra, MD, Study Chair — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Post Graduate institute Of Medical Education and Research, Chandigarh, Chandigarh, India